CLINICAL TRIAL: NCT03516474
Title: Minimally Disruptive Medicine: Reducing Treatment Burden and Improving Access for All Patients With Diabetes Using an mHealth Strategy
Brief Title: Using mHealth to Modernize Diabetes Care
Acronym: MDM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: South Riverdale Community Health Centre (Unknown); West Park Healthcare Centre (Other); Women's College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 17-365C
Record Dates: First submitted 2018-03-08; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Foot
Keywords: nir; diabetes; diabetic foot ulcer (DFU).; wound
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- St. Michael's Hospital: St. Michael's Hospital is an Acute care centre for the diabetic lower extremity.
  n=100
  Interventions: Device: MIMOSA Diagnostics
- South Riverdale Community Health Centre: South Riverdale is a Community Health Centre focused on prevention. n=100
  Interventions: Device: MIMOSA Diagnostics
- Westpark: Westpark is a rehabilitation site focused on post-operative/amputation care and preservation of the opposite limb. n=100
  Interventions: Device: MIMOSA Diagnostics
- Women's College Hospital: Women's College Hospital is an outpatient wound clinic focused on the management of DFUs. n=100
  Interventions: Device: MIMOSA Diagnostics

INTERVENTIONS:
Device: MIMOSA Diagnostics — The MIMOSA shines different "colours" of light on your skin. It will not touch your skin, or change how your wound is healing. The MIMOSA is designed to be used alongside the camera that is built into your cell phone, and we will use a cell phone to take a picture of your skin. This picture will tell us how much oxygen is getting to your wound, which can tell us more about how you are healing. The MIMOSA device is an experimental diagnostic tool, and will not influence how your wound is healing.
  Other Names: MIMOSA

SUMMARY:
In this study the investigators are testing a device that may help us tell how well the participants' wound is healing. This device is called the MIMOSA, and it shines different "colours" of light on the participants' skin. It will not touch the participants' skin, or change how the participants' wound is healing. The MIMOSA is designed to be used alongside the camera that is built into the participants' cell phone, and the investigators will use a cell phone to take a picture of the participants' skin. This picture will tell us how much oxygen is getting to the participants' wound, which can tell us more about how the participants are healing. The MIMOSA device is an experimental diagnostic tool, and will not influence how the participants' wound is healing.

DETAILED DESCRIPTION:
The investigators have developed a tool called the MultIspectral MObile TiSsue Assessment (MIMOSA) Device, which attaches to a smartphone and assesses tissue health parameters in a quick, non-invasive way using near-infrared light. This study will use MIMOSA to monitor patients at 4 sites in Toronto (St. Michael's Hospital, Women's College Hospital, South Riverdale Community Health Centre and at Westpark Healthcare Centre). These study sites were chosen to cover patients from diverse clinical backgrounds: St. Michael's Hospital is an Acute care centre for the diabetic lower extremity, Women's College Hospital is an outpatient wound clinic focused on the management of DFUs, South Riverdale is a Community Health Centre focused on prevention, and Westpark is a rehabilitation site focused on post-operative/amputation care and preservation of the opposite limb. conducted on patients who present with a non-healing diabetic foot ulcer and are already receiving standard best practice as prescribed by the diabetic foot multi-disciplinary team.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes: Type I or Type II.
2. Outpatient or inpatient
3. Diabetic Foot Ulcer
4. Adhere to monitoring schedule

Exclusion Criteria:

1. Presence of invasive infection requiring intravenous antibiotics
2. Cognitively able to give consent & participate in study
3. Active malignancy
4. End stage renal disease
5. Patients who are participating in another clinical study for ulcer management
6. Patients with a known history of poor compliance with medical treatment
7. Patients who are unable to understand the aims of the study and not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult diabetic subjects will be identified as candidates for our study if they present to the outpatient clinic, emergency department, inpatient or wound care team with or without a DFU. A subject is considered a patient with a DFU on one foot. If the patient has 2 wounds on the same foot, they are still considered one subject and both wounds are imaged. If the subject has a wound on the opposite foot they are considered a new subject.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower rates of DFU recurrence in patients monitored using mHealth | 0-12 months
  Accurately recorded pictures and information will help clinicians to accurately access patient foot health and hopefully reduce the frequency of DFU's using this information.

IPD SHARING:
Plan to Share IPD: No
All personal health information given will be anonymized when it is collected: a master linking log will link potentially identifiable characteristics to a specific study ID number listed in the app, to be held only by the Principal Investigator under lock or encryption and password protection. Study data seen by research assistants and data analysts will be strictly anonymized, encrypted, password protected, and stored in a locked research lab, separately from the master linking log.

REFERENCES:
- [Background] Pelletier C, Dai S, Roberts KC, Bienek A, Onysko J, Pelletier L. Report summary. Diabetes in Canada: facts and figures from a public health perspective. Chronic Dis Inj Can. 2012 Dec;33(1):53-4. PMID 23294922
- [Background] Skrepnek GH, Mills JL Sr, Armstrong DG. A Diabetic Emergency One Million Feet Long: Disparities and Burdens of Illness among Diabetic Foot Ulcer Cases within Emergency Departments in the United States, 2006-2010. PLoS One. 2015 Aug 6;10(8):e0134914. doi: 10.1371/journal.pone.0134914. eCollection 2015. PMID 26248037
- [Background] Serrano V, Spencer-Bonilla G, Boehmer KR, Montori VM. Minimally Disruptive Medicine for Patients with Diabetes. Curr Diab Rep. 2017 Sep 23;17(11):104. doi: 10.1007/s11892-017-0935-7. PMID 28942581
- [Background] Cross KM, Leonardi L, Payette JR, Gomez M, Levasseur MA, Schattka BJ, Sowa MG, Fish JS. Clinical utilization of near-infrared spectroscopy devices for burn depth assessment. Wound Repair Regen. 2007 May-Jun;15(3):332-40. doi: 10.1111/j.1524-475X.2007.00235.x. PMID 17537120
- [Background] Vashist SK, Schneider EM, Luong JH. Commercial Smartphone-Based Devices and Smart Applications for Personalized Healthcare Monitoring and Management. Diagnostics (Basel). 2014 Aug 18;4(3):104-28. doi: 10.3390/diagnostics4030104. PMID 26852680